CLINICAL TRIAL: NCT06465199
Title: A Dose Escalation Study Using Eflornithine (DFMO) and AMXT 1501 Followed by a Randomized Controlled Trial of DFMO With or Without AMXT 1501 for Neuroblastoma, CNS Tumors, and Sarcomas
Brief Title: Eflornithine (DFMO) and AMXT 1501 for Neuroblastoma, CNS Tumors, and Sarcomas
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Aminex Therapeutics, Inc. (Industry); Penn State University (Other)
Responsible Party: Principal Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BCC020
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Atypical Teratoid/Rhabdoid Tumor; Embryonal Tumor With Multilayered Rosettes; Ewing Sarcoma; Diffuse Intrinsic Pontine Glioma; Osteosarcoma; Neuroblastoma
MeSH Terms: conditions — Rhabdoid Tumor; Neuroectodermal Tumors, Primitive; Sarcoma, Ewing; Diffuse Intrinsic Pontine Glioma; Osteosarcoma; Neuroblastoma | interventions — Eflornithine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I- AYA Cohort (Experimental): The initial phase I will be an AYA (adolescents and young adult) cohort that will be for subjects ≥12 years of age at enrollment in a standard 3+3 design in which groups of 3 subjects per cohort will be treated and assessed. Subjects will receive up to twenty-four (24), 28-day cycles of AMXT 1501 combined with DFMO. Subjects will receive oral AMXT 1501 at a starting dose of 350 mg/m2 BID each day. The dose escalation scheme for subsequent groups and modifications for dose limiting toxicities (DLT) are detailed in the protocol.
  Interventions: Drug: Eflornithine (DFMO); Drug: AMXT 1501 Dicaprate
- Phase I- Pediatric Cohort (Experimental): The second phase I will be a pediatric cohort that will be for subjects < 12 years of age at enrollment in a standard 3+3 design in which groups of 3 subjects per cohort will be treated and assessed. Subjects will receive up to twenty-four (24), 28-day cycles of AMXT 1501 combined with DFMO. Subjects will receive oral AMXT 1501 at a starting dose of 350 mg/m2 BID each day. The dose escalation scheme for subsequent groups and modifications for dose limiting toxicities (DLT) are detailed in the protocol.
  Interventions: Drug: Eflornithine (DFMO); Drug: AMXT 1501 Dicaprate
- Phase II- Arm A: AMXT 1501 + DFMO (Experimental): In this portion of the study, cohort 1 will be randomized to either receive Arm A: oral AMXT 1501 at the recommended phase 2 dose (RP2D) found in the Phase I along with oral DFMO at the RP2D found in the Phase I on each day of study or Arm B: oral DFMO alone at the recommended phase 2 dose (RP2D) found in the Phase I. Subjects will receive up to twenty-four (24), 28-day cycles of their assigned treatment. Cohorts 2 (ETMR/ATRT), 3 (DIPG), and 4 (Sarcomas) will automatically be assigned to Arm A with AMXT 1501 in combination with DFMO.
  Subjects in cohort 1 who progress on DFMO alone (and have met the primary PFS endpoint) may cross over to AMXT 1501+DFMO.
  Interventions: Drug: Eflornithine (DFMO); Drug: AMXT 1501 Dicaprate
- Phase II- Arm B: DFMO Alone (Active Comparator): In this portion of the study, cohort 1 will be randomized to either receive Arm A: oral AMXT 1501 at the recommended phase 2 dose (RP2D) found in the Phase I along with oral DFMO at the RP2D found in the Phase I on each day of study or Arm B: oral DFMO alone at the recommended phase 2 dose (RP2D) found in the Phase I. Subjects will receive up to twenty-four (24), 28-day cycles of their assigned treatment. Cohorts 2 (ETMR/ATRT), 3 (DIPG), and 4 (Sarcomas) will automatically be assigned to Arm A with AMXT 1501 in combination with DFMO.
  Subjects in cohort 1 who progress on DFMO alone (and have met the primary PFS endpoint) may cross over to AMXT 1501+DFMO.
  Interventions: Drug: Eflornithine (DFMO)

INTERVENTIONS:
Drug: Eflornithine (DFMO) — Oral DFMO capsules
  Other Names: Difluoromethylornithine
Drug: AMXT 1501 Dicaprate — Capsule
  Arms: Phase I- AYA Cohort; Phase I- Pediatric Cohort; Phase II- Arm A: AMXT 1501 + DFMO

SUMMARY:
The purpose of this study is to evaluate the investigational oral drug AMXT 1501 in combination with oral eflornithine (DFMO). An investigational drug is one that has not been approved by the U.S. Food & Drug Administration (FDA), or any other regulatory authorities around the world for use alone or in combination with any drug, for the condition or illness it is being used to treat.

The goals of this part of the study are:

* Establish a recommended dose of AMXT 1501 in combination with DFMO
* Test the safety and tolerability of AMXT 1501 in combination with DFMO
* To determine the activity of study treatments chosen based on:
* How each subject responds to the study treatment
* How long a subject lives without their disease returning/progressing

ELIGIBILITY:
Inclusion Criteria:

1. Age:

   All subjects: Must be a maximum of 21 years of age at diagnosis

   Age at enrollment by Phase:
   1. Phase I-AYA (adolescents and young adult) Cohort: ≥12 years of age at enrollment.
   2. Phase I-Pediatric Cohort: < 12 years of age at enrollment; may start only after DSMB review confirms the RP2D from the AYA cohort. No subject < 12 years will be treated at a dose level higher than the RP2D established in the Phase I-AYA Cohort.
   3. Phase II: ≤ 21 years of age at diagnosis (with possibly two different age-specific RP2Ds).
2. Pathology

   All subjects must have a confirmed pathologic diagnosis of tumor type (except for DIPG):
   * Relapsed/refractory Neuroblastoma (NB)
   * Relapsed/refractory Embryonal tumor with multilayer rosettes (ETMR)
   * Relapsed/refractory Atypical teratoid rhabdoid tumor (ATRT)
   * Newly diagnosed Diffuse Intrinsic Pontine Glioma (DIPG)- radiologic diagnosis acceptable
   * Relapsed/refractory Ewing Sarcoma (EWS)
   * Relapsed/refractory Osteosarcoma (OST)
3. Tumor assessment:

   Disease staging must be performed at baseline during the 28 day screening period prior to first dose of study drug.
4. Disease Status:

   Relapsed or Refractory Neuroblastoma Relapsed disease defined as: High-risk neuroblastoma that was previously in remission after standard therapy (at least 4 cycles of aggressive multi-drug induction chemotherapy, with or without radiation, surgery, and immunotherapy, or according to a standard high-risk treatment/neuroblastoma protocol).

   Refractory disease defined as: High-risk neuroblastoma that 1) failed to achieve CR after at least 4 cycles of aggressive multi-drug induction chemotherapy with or without radiation and surgery, followed by immunotherapy, or according to a standard high-risk treatment/neuroblastoma protocol, or 2) progression during upfront therapy or 3) with disease remaining after standard immunotherapy.

   Eligible NB subjects may have active disease or no active disease.

   NB Subjects with no active disease need to meet the following criteria:

   Timing from prior therapy: Enrollment (first dose of study drug) no later than 60 days from most recent therapy.

   NB Subjects with active disease need to meet the following criteria:
   * Received at least one recent treatment for their relapse/refractory disease and is stable (SD) or better on this treatment.

     *Stable disease defined as non-progression over 2 separate imaging studies at least 6 weeks apart
   * Subjects must not have disease in any organs (including lungs, liver, or brain).
   * Measurable tumor size is < 2 cm
   * Bone marrow < 40% involvement

   Relapsed or refractory ETMR/ATRT Subjects that have relapsed following standard of care therapy or having progressed during standard of care therapy and non-responsive/progressive to accepted curative therapy, including up-front chemotherapy and radiation and/or high-dose chemotherapy with stem cell rescue.

   ETMR/ATRT Subjects with no active disease need to meet the following criteria:

   Timing from prior therapy: Enrollment (first dose of study drug) no later than 60 days from most recent therapy.

   ETMR/ATRT Subjects with active disease need to meet the following criteria:

   • Received at least one recent treatment for their relapse/refractory disease and is stable (SD) or better on this treatment.

   *Stable disease defined as non-progression over 2 separate imaging studies at least 6 weeks apart

   Newly Diagnosed Diffuse Intrinsic Pontine Glioma (DIPG) Subjects with DIPG to start greater than 30 days, and no longer than 60 days, after standard of care radiation therapy.

   Subjects with newly-diagnosed typical DIPG, defined as tumors with a pontine epicenter and diffuse involvement of the pons on at least 1 axial T2-weighted image, are eligible. No histologic confirmation is required. Subjects with metastatic disease are not eligible. Subjects with a biopsy and no evidence of H3K27m mutations are eligible as long as they meet radiographic criteria. Subjects with H3K27m altered DMG outside of the brainstem are not eligible. Subjects with progression or recurrence after initial standard of care radiation are ineligible.

   Relapsed or refractory Ewing sarcoma and osteosarcoma Subjects that have relapsed following standard of care therapy or having progressed during standard of care therapy. Standard of care therapy for Ewing sarcoma and osteosarcoma includes multi-agent chemotherapy with local control consisting of either surgery or radiation therapy.

   EWS/OST Subjects with no active disease need to meet the following criteria:

   Timing from prior therapy: Enrollment (first dose of study drug) no later than 60 days from most recent therapy.

   EWS/OST Subjects with active disease need to meet the following criteria:

   • Received at least one recent treatment for their relapse/refractory disease and is stable (SD) or better on this treatment.

   *Stable disease defined as non-progression over 2 separate imaging studies at least 6 weeks apart
5. Subjects must be able to swallow capsules.
6. Subjects with CNS disease currently taking steroids must have been on a stable dose of steroids for at least one week and must not have progressive hydrocephalus at enrollment.
7. Subjects must have fully recovered from the acute toxic effects of all prior anti- cancer chemotherapy and be within the following timelines:

   1. Myelosuppressive chemotherapy: Must not have received within 2 weeks of enrollment onto this study (6 weeks if prior nitrosourea).
   2. Small Molecule Inhibitor (anti-neoplastic agent): At least 7 days since the completion of therapy with a small molecule inhibitor. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the Study Chair.
   3. Immunotherapy: At least 4 weeks since the completion of any type of immunotherapy, e.g. tumor vaccines, CAR-T cells except for anti-GD2 Monoclonal antibodies (ex. naxitamab, dinutuximab, etc.) which should be at least 2 weeks since prior treatment with a monoclonal antibody.
   4. XRT: At least 14 days since the last treatment except for radiation delivered with palliative intent to a non-target site.

      Note: Subjects with DIPG will be required to have had up front standard of care radiation. As above, subjects with DIPG must be between 30-60 days post initial up front radiation therapy.
   5. Stem Cell Transplant:

      1. Allogeneic: No evidence of active graft vs. host disease
      2. Allo/Auto: ≥ 45 days must have elapsed since transplant.
   6. MIBG Therapy: At least 6 weeks since treatment with MIBG therapy.
8. Subjects must have a Lansky or Karnofsky Performance Scale score of >/= 60
9. Subjects must have adequate organ function at the time of enrollment:

   * Hematological: Hematological recovery as defined by ANC ≥750/μL (unsupported- >24 hrs off G-CSF and 7 days off neulasta)
   * Liver: Adequate liver function as defined by AST and ALT <10x upper limit of normal
   * Cardiac: all subjects must have:

     1. Normal serum Cardiac Troponin Concentration
     2. Normal BNP (B-type natriuretic peptide) Level
     3. A QTcF ≤ 470 msec (or EKG with no significant findings)
     4. Normal ECHO defined as:

     i. Shortening fraction of ≥ 27% by echocardiogram, or ii. Ejection fraction of ≥ 50% by echocardiogram or radionuclide angiogram
   * Renal: Subjects must have adequate renal function defined as:

     1. For subjects < 17 years old: estimated Glomerular Filtration rate (eGFR) as calculated from the Bedside Schwartz equation (in units of mL/min/1.73 m2) or via radioisotope GFR of ≥ 70 mL/min/1.73 m2. The Bedside Schwartz equation is: [(0.413) X (Height in cm)] / SCr
     2. For subjects ≥17 years old: estimated Glomerular Filtration rate (eGFR) as calculated from the Cockcroft and Gault formula (in units of mL/min/1.73 m2) or via radioisotope GFR of ≥ 70 mL/min/1.73 m2. The Cockcroft and Gault formula is: [(140-age) x (Wt in kg) x (0.85 if female)] / (72 x SCr)
     3. OR a 24 hour urine Creatinine clearance ≥ 70 mL/min/1.73 m2
10. Subjects of childbearing potential must have a negative pregnancy test. Subjects of childbearing potential must agree to use an effective birth control method. Subjects who are lactating must agree to stop breast-feeding.
11. Written informed consent in accordance with institutional and FDA guidelines must be obtained from all subjects (or subjects' legal representative).

Exclusion Criteria:

1. BSA of <0.25 m2
2. Investigational Drugs: Subjects who are currently receiving another investigational drug are excluded from participation.
3. Anti-cancer Agents: Subjects who are currently receiving other anticancer agents are not eligible. Subjects must have fully recovered from the hematological and bone marrow suppression effects of prior chemotherapy.
4. Infection: Subjects who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
5. Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 289 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2033-02 (Estimated); Study Completion 2035-02 (Estimated)

PRIMARY OUTCOMES:
Phase I- Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 28 days
  To evaluate the safety, tolerability and recommended phase 2 dose (RP2D) of AMXT 1501 in combination with oral DFMO in pediatric and young adult subjects.
Phase II- Number of Cohort 1 participants with progression free survival (PFS) during study | 2 years plus 5 years follow up
  To evaluate, in a prospective randomized clinical trial, the efficacy of eflornithine (DFMO) in combination with AMXT 1501 compared to DFMO alone in neuroblastoma (Cohort 1) based upon Progression Free Survival (PFS)
Phase II- Number of Cohort 2-4 participants with progression free survival (PFS) during study | 2 years plus 5 years follow up
  To evaluate the efficacy of eflornithine (DFMO) in combination with AMXT 1501 in non-randomized (Cohorts 2-4) based upon Progression Free Survival (PFS):
  2. Cohort 2-Relapsed/refractory Embryonal Tumor with Multilayered Rosettes (ETMR) Atypical Teratoid Rhabdoid Tumor (ATRT) 3. Cohort 3-Diffuse Intrinsic Pontine Glioma (DIPG) at diagnosis after standard of care radiation therapy 4. Cohort 4- Relapsed/refractory Ewing Sarcoma (EWS) and Osteosarcoma (OST)

SECONDARY OUTCOMES:
Phase I- Number of participants with progression free survival (PFS) during study | 2 years plus 5 years follow up
  To evaluate the activity of AMXT 1501 in combination with DFMO based on Progression free survival (PFS)
Phase I- Determine the Overall Response Rate (ORR) of Participants using INSS Response | 2 years
  To evaluate the activity of AMXT 1501 in combination with DFMO based on Overall response rate (ORR)
Phase II- Determine the Overall Response Rate (ORR) of Participants using INSS Response | 2 years
  To evaluate the efficacy of eflornithine (DFMO) in combination with AMXT 1501 (Cohort 2-4) and in a randomized arm compared to DFMO alone in neuroblastoma (Cohort 1), based upon overall response rate (ORR).
Phase II- Length of time that participants experience Overall Survival (OS) | 2 years plus 5 years follow up
  To evaluate the efficacy of eflornithine (DFMO) in combination with AMXT 1501 (Cohort 2-4) and in a randomized arm compared to DFMO alone in neuroblastoma (Cohort 1), based upon overall Survival (OS).
Phase II-Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years plus 30 days
  To evaluate the safety and tolerability profile of eflornithine (DFMO) in combination with AMXT 1501 in pediatric and young adult subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Saulnier Sholler, MD, Study Chair — Penn State Health Children's Hospital
Locations (4):
- United States (4):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Connecticut Children's Hospital, Hartford, Connecticut
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Beat Childhood Cancer Research Consortium website — https://research.beatcc.org/